CLINICAL TRIAL: NCT04378582
Title: Characteristics and Outcomes of Patients With COVID-19 Admitted to the ICU
Acronym: EpiCoV-Brazil
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Juliana Carvalho Ferreira, Assistant professor, University of Sao Paulo General Hospital
Other Study IDs: 31382620.0.0000.0068
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: SARS-CoV 2; Respiratory Distress Syndrome, Adult; Corona Virus Infection; Critical Illness
Keywords: Critical Care
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections; Critical Illness | interventions — Risk Factors; Demography; Comorbidity; Health Services Needs and Demand

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 confirmed: Patients with confirmed COVID-19 by RT-PCR or serological test
  Interventions: Other: risk factors
- COVID-19 suspected: Patients suspected COVID-19, as defined by clinical history and course, who have negative RT-PCR or serological test but where treated and cared for as COVID-19 patients
  Interventions: Other: risk factors

INTERVENTIONS:
Other: risk factors — This is an observational study, so there are no interventions. Investigators will collect data about demographics, comorbidities, and other risk factors such as severity of disease at admission, need for advanced life support, need for invasive mechanical ventilation and ventilator parameters on day1 of mechanical ventilation or ICU admission as potentially association with survival
  Other Names: demographics; comorbidities; mechanical ventilation parameters; need for advanced life support

SUMMARY:
This is a case series of patients with COVID-19 admitted to the largest university hospital in Sao Paulo, Brazil, during the 2020 COVID-19 pandemic. Data will be collected prospectively and retrospectively.

The main objective is to describe the characteristics of critically ill patients with COVID-19 and their clinical outcomes, and to identify risk factors associated with survival, to inform clinical decision-making and to guide the strategy to mitigate the epidemic, both within each hospital and ICU and in public health management.

DETAILED DESCRIPTION:
In December 2019, an outbreak of Severe Acute Respiratory Syndrome (SARS) attributed to a new coronavirus, called SARS-CoV-2, was described in the Wuhan region of China. This SARS, caused by SARS-CoV-2 was called COVID-19, spread across the globe, causing millions of cases on all continents, and thousands of deaths, being characterized as a pandemic.

COVID-19 is characterized by a flu-like syndrome, with symptoms such as fever, cough, myalgia and gastrointestinal symptoms. Most cases are mild, some even asymptomatic, but approximately 15% of patients have more severe presentation, and approximately 5% are critical (7).

The acute respiratory failure of critically ill patients with COVID-19 has different aspects, including hypoxemia of difficult treatment, associated in some cases with clotting disorders, changes in immunity and inflammatory phenomena that pose challenges for the management of these patients, whose mortality can be high.

The Hospital das Clínicas da Faculdade de Medicina de São Paulo implemented an action plan that provides for the creation of 200 ICU beds to serve patients with COVID-19. Knowing the characteristics of critically ill patients with COVID-19 and their clinical outcomes is extremely important to inform clinical decision-making and to guide the strategy to mitigate the epidemic, both within each hospital and ICU and in public health management.

ELIGIBILITY:
Inclusion Criteria:

* Being admitted to one of the COVID-19 ICUs during the study period
* Suspected or confirmed COVID-19
* Expected ICU stay greater than 24 hours

Exclusion Criteria:

* ICU Readmission during the same hospital stay (patients will be evaluated only during their first ICU stay)

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed COVID-19 by RT-PCR or sorological test, or suspected COVID-19, as defined by clinical history and course, who have negative RT-PCR or sorological test but where treated and cared for as COVID-19 patients, who are admitted to the ICU during the study period.
  Data will be collected prospectively for patients admitted to the ICU after the the date of study approval and retrospectively for patients admitted to the ICU during the COVID-19 epidemic in sao paulo, but before the study was initiated.
  A sample size of 300 patients was inittialy anticipated. As the epidemic in Sao Paulo grew fast, the hospital opened new ICU beds and the investigators reviewed the anticipated sample size to 500 patients. Given that the study has no risks for participants, and that informed consent was waived by the IRB, investigators intend to collect data about all patients with COVID-19 admitted to the ICUs during the study period, possibly more than the anticipated sample size.
Sampling Method: Non-Probability Sample
Enrollment: 1589 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
ICU survival at 28 days | 28 days
  the proportion of patients who survive to ICU discharge or for 28 days in the ICU

SECONDARY OUTCOMES:
Hospital survival at 60 days | 60 days
  the proportion of patients who survive to hospital discharge or for 60 days in the hospital
Duration of mechanical ventilation | 28 days
  Number of days under invasive ventilatory support
Need for renal replacement therapy | 28 days
  Proportion of patients who received renal replacement therapy during the ICU stay
Complications during the ICU stay | 28 days
  percentage of patients who developed complications during the ICU stay: thromboembolic events, ventilator associated pneumonia, secondary infections, cardiovascular complications

CONTACTS AND LOCATIONS:
Overall Officials: Juliana C Ferreira, MD, Principal Investigator — University of Sao Paulo - hospital das Clínicas da faculdade de medicina da USP (HCFMUSP)
Locations (1):
- Hospital das Clínicas -HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The investigators haven't developed a plan for sharing, but would be open to share unidentified data for research or public health purposes

REFERENCES:
- [Derived] Taniguchi LU, Aliberti MJR, Dias MB, Jacob-Filho W, Avelino-Silva TJ. Calculating Route: Functional Trajectories and Long-Term Outcomes in Survivors of Severe COVID-19. J Nutr Health Aging. 2023;27(12):1168-1173. doi: 10.1007/s12603-023-2036-4. PMID 38151867
- [Derived] Taniguchi LU, Avelino-Silva TJ, Dias MB, Jacob-Filho W, Aliberti MJR; COVID-19 and Frailty (CO-FRAIL) Study Group and EPIdemiology of Critical COVID-19 (EPICCoV) Study Group, for COVID Hospital das Clinicas, University of Sao Paulo Medical School (HCFMUSP) Study Group. Patient-Centered Outcomes Following COVID-19: Frailty and Disability Transitions in Critical Care Survivors. Crit Care Med. 2022 Jun 1;50(6):955-963. doi: 10.1097/CCM.0000000000005488. Epub 2022 Jan 26. PMID 35081061
- [Derived] Ferreira JC, Ho YL, Besen BAMP, Malbuisson LMS, Taniguchi LU, Mendes PV, Costa ELV, Park M, Daltro-Oliveira R, Roepke RML, Silva JM Jr, Carmona MJC, Carvalho CRR; EPICCoV Study Group; Hirota A, Kanasiro AK, Crescenzi A, Fernandes AC, Miethke-Morais A, Bellintani AP, Canasiro AR, Carneiro BV, Zanbon BK, Batista BPSN, Nicolao BR, Besen BAMP, Biselli B, Macedo BR, Toledo CMG, Pompilio CE, Carvalho CRR, Mol CG, Stipanich C, Bueno CG, Garzillo C, Tanaka C, Forte DN, Joelsons D, Robira D, Costa ELV, Silva EM Junior, Regalio FA, Segura GC, Marcelino GB, Louro GS, Ho YL, Ferreira IA, Gois JO, Silva JM Junior, Reusing JO Junior, Ribeiro JF, Ferreira JC, Galleti KV, Silva KR, Isensee LP, Oliveira LS, Taniguchi LU, Letaif LS, Lima LT, Park LY, Chaves L Netto, Nobrega LC, Haddad L, Hajjar L, Malbouisson LM, Pandolfi MCA, Park M, Carmona MJC, Andrade MCPH, Santos MM, Bateloche MP, Suiama MA, Oliveira MF, Sousa ML, Louvaes M, Huemer N, Mendes P, Lins PRG, Santos PG, Moreira PFP, Guazzelli RM, Reis RB, Oliveira RD, Roepke RML, Pedro RAM, Kondo R, Rached SZ, Fonseca SRS, Borges TS, Ferreira T, Cobello V Junior, Sales VVT, Ferreira WSC. Characteristics and outcomes of patients with COVID-19 admitted to the ICU in a university hospital in Sao Paulo, Brazil - study protocol. Clinics (Sao Paulo). 2020;75:e2294. doi: 10.6061/clinics/2020/e2294. Epub 2020 Aug 26. PMID 32876113